CLINICAL TRIAL: NCT02861911
Title: Effects of NMES on Muscle Function of Patients With FSHD: a Double-blind Randomized Controlled Clinical Trial
Brief Title: Effects of NMES on Muscle Function of Patients With FSHD: a Double-blind Randomized Controled Clinical Trial
Acronym: NEMS and FSHD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty in recruiting patients
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: UF 9344
Record Dates: First submitted 2016-08-03; First posted 2016-08-10 (Estimated); Last update posted 2019-05-09 (Actual); Status verified 2019-05

CONDITIONS: Primary Disease Facioscapulohumeral Dystrophy (FSHD)
Keywords: Muscle function; Oxidative stress; Quality of life; Physical activities
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (Sham Comparator): The current intensity is generally defined between the sensory and motor threshold (patients feel the power but no visible muscle contraction will be obtained).
  Interventions: Other: Current flow between sensory and motor threshold
- Active NMES group (Active Comparator): Tthe current intensity must always meet and exceed the motor threshold (patients feel the current and quadriceps muscle will contract a visible and quantifiable if possible).
  Interventions: Device: Current intensity upper of motor threshold by Kneehab XP technology

INTERVENTIONS:
Other: Current flow between sensory and motor threshold — Artificial strength training by means of neuromuscular electrical stimulation (NMES)
  Arms: Control group
Device: Current intensity upper of motor threshold by Kneehab XP technology — Artificial strength training by means of neuromuscular electrical stimulation (NMES)
  Arms: Active NMES group

SUMMARY:
Facioscapulohumeral muscular dystrophy (FSHD) is an autosomal dominant disease characterized by progressive weakness and atrophy of specific skeletal muscles. One of the major problems of patients affected by FSHD is the limitation in performing daily activities induced by the progressive muscle weakness. This sedentary lifestyle can cause a "debilitative cycle," and neuromuscular deconditioning can even aggravate the muscular deficiencies. Recent studies have indicated the safety and the effectiveness of moderate aerobic training programs in patients with FSHD. However, these training programs have limited applicability in patients with more severe muscular weakness. Artificial strength training by means of neuromuscular electrical stimulation (NMES) appears to be a promising rehabilitation strategy for FSHD patients suffering from neuromuscular disorders. Therefore we propose to investigate the feasibility, safety, and effectiveness of NMES strength training to counteract quadriceps muscle weakness in patients affected by FSHD.

DETAILED DESCRIPTION:
NMES will be delivered to both quadriceps by means of a Kneehab® XP device, which is an innovative and clinically-proven garment-based product designed specifically to treat quadriceps muscle atrophy. The main NMES current parameters are: 50-Hz frequency, 100-400 µs pulse duration, 5:10-second on:off time. Each session will last approximately 20 minutes and will be repeated 5 days/week for a total duration of the treatment program of 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Molecular and/or clinical diagnosis for FSHD
* Vignos scale ≤ 5: Able to walk without help
* Clinically characterized by quadriceps muscle weakness but with a maximal voluntary contraction (MVC) between 8 and 16 Kg
* Follow as part of their usual care in the Clinical Physiology Department of the University Hospital of Montpellier
* Free and informed consent of the patient
* Patient affiliated or beneficiary of a social security system

Exclusion Criteria:

* Patient with co-morbidity:pathologies heart, pathologies respiratory, metabolic and endocrine -pathologies, pathologies cancer.
* Patients treated with drugs could cause muscle side effects or interfere with muscle metabolism.
* Lesions or skin inflammation at the thighs that can prevent the application of NMES
* Claustrophobic subject
* Carrier of intracranial vascular clip, cardiac pacemaker, neurostimulator, cochlear implant, or intraocular metallic foreign
* Pregnant or nursing women
* Vulnerable Persons and protected Major or unable to consent
* Patient in exclusion period relative over another protocol, or for which the annual amount of maximum compensation of € 4,500 has been reached

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2015-10-20 (Actual); Primary Completion 2016-09-13 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Maximal voluntary contraction (MVC) strength of the quadriceps | At 3 months

SECONDARY OUTCOMES:
Effect of NEMS on the quality of life (SF36 questionnaire) | At 3 months
Effect of NMES on the quadriceps endurance evaluated in a dynamic test against a charge equal to 30% of maximal isometric force. | At 3 months
Evaluation of the body composition by bioelectric impedance analysis (BIA) after NMES effect | At 3 months
Effect of NMES on the bone mineral density by dual energy X-ray absorptiometry (DEXA) | At 3 months
Effect of NMES on the oxidative stress markers in blood and urine by blood and urine tests | At 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Montpellier University Hospital, Montpellier, France